CLINICAL TRIAL: NCT07056907
Title: Evaluating the Neuroprotective Effects of Continuous Lumbar Drainage on the Cerebral Perfusion in Patients With an Acute Ischemic Stroke and Hemodynamic Failure Type 2: a Pilot Study
Brief Title: Effects of Cerebrospinal Fluid Drainage on Cerebral Hemodynamics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Christiaan van Niftrik, Dr. sc. med., University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INOV00181
Record Dates: First submitted 2025-06-18; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Acute Ischemic Stroke
Keywords: BOLD-CVR; fMRI; lumbar drain; stroke; acute; ischemia; large vessel occlusion
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label, prospective interventional study in which all participants receive the same intervention: temporary cerebrospinal fluid (CSF) drainage via lumbar drain. Each participant serves as their own control, with pre- and post-intervention imaging used to assess within-subject changes in cerebrovascular reactivity (CVR), as measured by BOLD-CVR MRI.
  There is no randomization or blinding. This design is appropriate for an early-phase, mechanistic pilot trial aiming to determine physiological feasibility, safety, and proof-of-concept effect of the intervention.
  To provide context for naturally occurring temporal changes in BOLD-CVR, outcomes will be compared to a matched historical control cohort of acute ischemic stroke patients who underwent serial BOLD-CVR imaging without any intervention. This external comparison is not considered a formal control arm but supports exploratory evaluation of treatment-related effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumbar Drainage in Acute Ischemic Stroke Patients With Hemodynamic Failure (Single Intervention Arm) (Experimental): Patients with acute ischemic stroke and evidence of hemodynamic failure on BOLD-CVR MRI (hemispheric CVR ≤ 0.1041 or MCA territory CVR ≤ 0.0778) will receive temporary cerebrospinal fluid (CSF) drainage via a lumbar drain. The drain will be placed under sterile conditions by experienced neurosurgical staff and connected to a closed CSF drainage system. Continuous drainage will be performed for approximately 48 to 72 hours under standardized pressure-controlled conditions. Each patient undergoes BOLD-CVR MRI before and after the drainage period to assess changes in cerebrovascular reactivity. Clinical outcomes (NIHSS, mRS) and safety events (e.g., infection, CSF leak) will also be recorded. This arm is open-label and includes only a single group receiving the intervention.
  Interventions: Procedure: Lumbar drain placement

INTERVENTIONS:
Procedure: Lumbar drain placement — This intervention involves temporary cerebrospinal fluid (CSF) drainage via lumbar drain in acute ischemic stroke patients with MRI-confirmed hemodynamic failure. The lumbar drain is inserted at the bedside or in a procedural suite under sterile conditions and connected to a pressure-regulated, closed drainage system. Drainage is continuous for 48-72 hours, with volume and pressure carefully monitored. This intervention is distinct in targeting stroke patients without hydrocephalus, using CSF drainage as a novel method to improve cerebral perfusion and vascular reserve. The effect is evaluated with serial BOLD-CVR MRI performed before and after the drainage period, making this one of the first interventional stroke studies to use functional MRI as a physiological endpoint.

SUMMARY:
This pilot interventional study investigates whether continuous cerebrospinal fluid (CSF) drainage via lumbar drain can improve cerebrovascular reactivity (CVR) in patients with acute ischemic stroke and hemodynamic failure, as assessed by blood oxygenation level dependent (BOLD) MRI.

Patients with acute ischemic stroke frequently exhibit impaired cerebral autoregulation and reduced vascular reserve. In such cases, a low BOLD-CVR response is associated with a high (~40%) risk of recurrent ischemic stroke despite optimal medical therapy. Hemodynamic failure stage 2 (HF2), defined by severely reduced CVR (hemispheric BOLD-CVR ≤ 0.1041), indicates exhausted compensatory capacity and poor perfusion.

Evidence from other neurological conditions suggests that CSF drainage via lumbar drain may transiently lower intracranial pressure, improve perfusion, and enhance autoregulatory function. This study aims to apply these findings to acute stroke patients with hemodynamic compromise.

Eligible patients will undergo BOLD-CVR MRI to assess cerebrovascular reserve. Those meeting HF2 criteria and without contraindications will be offered inclusion. After informed consent (or proxy consent), a lumbar drain will be placed, and continuous CSF drainage performed over ~48 hours. A follow-up BOLD-CVR MRI will assess changes in CVR. In addition, 20 ml of CSF will be extracted to evaluate acute effects on CVR. A historical cohort will be used to control for spontaneous CVR variation over 48 hours.

Primary Objective:

To determine whether continuous CSF drainage improves BOLD-CVR in patients with HF2 following acute ischemic stroke.

Secondary Objectives:

To compare longitudinal BOLD-CVR changes to a historical cohort. To evaluate safety and feasibility of lumbar drainage in this setting. To assess short-term clinical outcomes (NIHSS, mRS) and recurrent events. To assess BOLD-CVR change after 20 ml CSF extraction.

Study Design:

Single-center, open-label, prospective pilot study. Participants serve as their own control, with pre- and post-intervention imaging to evaluate physiological effects. Safety and exploratory clinical data will also be collected.

This proof-of-concept trial aims to generate preliminary evidence for a potential therapeutic strategy in high-risk stroke patients with poor autoregulation. Positive findings could inform future randomized controlled trials.

DETAILED DESCRIPTION:
This pilot interventional study explores the physiological and clinical impact of continuous cerebrospinal fluid (CSF) drainage via lumbar drain on cerebrovascular reactivity (CVR) in patients with acute ischemic stroke who exhibit hemodynamic failure, as measured by blood oxygenation level-dependent (BOLD) functional MRI.

Background and Rationale In patients with acute ischemic stroke, failure of autoregulatory capacity and exhaustion of cerebrovascular reserve represent major contributors to secondary ischemic injury and poor outcomes. Despite optimal medical management, patients with documented hemodynamic failure remain at high risk for recurrent ischemic stroke, often exceeding 30-40% within the first months post-event.

BOLD-CVR is a non-invasive MRI-based technique that maps the cerebrovascular response to a vasodilatory stimulus (commonly CO₂ or breath-hold induced hypercapnia). When interpreted using standardized processing pipelines, it offers a quantitative assessment of cerebral hemodynamics and can differentiate between regions with preserved, reduced, or exhausted vascular reserve. In previous research, a hemispheric mean BOLD-CVR ≤ 0.1041 or a middle cerebral artery (MCA) territory mean BOLD-CVR ≤ 0.0778 has been associated with hemodynamic failure stage 2 (HF2).

There is preliminary evidence from other neurological conditions (e.g., idiopathic intracranial hypertension, traumatic brain injury, and subarachnoid hemorrhage) that CSF diversion through lumbar drainage can lead to improved cerebral perfusion and functional outcomes. The proposed mechanism involves a transient reduction in intracranial pressure (ICP), improved compliance, and favorable shifts in cerebral perfusion pressure gradients. However, this strategy has not been evaluated in the context of acute ischemic stroke in patients without hydrocephalus but with severe autoregulatory impairment.

This study hypothesizes that temporary CSF drainage in such patients will improve BOLD-CVR as an imaging marker of vascular reserve and possibly influence clinical outcomes.

Study Objectives

Primary Objective:

To assess whether continuous CSF drainage via lumbar drain results in measurable improvement of cerebrovascular reactivity (BOLD-CVR) in acute ischemic stroke patients with HF2.

Secondary Objectives:

To evaluate the safety and technical feasibility of lumbar drain placement in acute stroke patients without hydrocephalus.

To explore changes in neurological function (NIH Stroke Scale and modified Rankin Scale) at discharge and during follow-up.

To monitor for recurrent ischemic stroke events during the subacute period post-intervention.

To compare observed CVR changes with those occurring naturally over time in a historical cohort with matched inclusion criteria but no CSF drainage.

Study Design and Methodology This is a prospective, single-center, open-label, pilot interventional trial. Patients admitted with acute ischemic stroke will undergo BOLD-CVR MRI within a defined time window (typically within 3-7 days post-event) to assess cerebrovascular reserve.

Inclusion criteria require radiologically confirmed acute ischemic stroke and a BOLD-CVR profile consistent with HF2. Patients with hydrocephalus, mass effect, active CNS infection, or contraindications to lumbar puncture are excluded.

Intervention: Eligible and consenting patients will undergo placement of a lumbar drain by experienced neurosurgical staff. Continuous drainage will be performed over a period of 48-72 hours using a pressure-controlled closed CSF system. Drainage volumes and pressures will be recorded in standardized templates.

Imaging Protocol: BOLD-CVR imaging will be performed at two time points:

Baseline scan: prior to lumbar drainage.

Follow-up scan: 12-24 hours after completion of drainage.

All imaging will be performed on the same scanner with identical acquisition parameters and stimulus paradigm (e.g., breath-hold or fixed hypercapnic challenge with end-tidal CO₂ monitoring). Data will be processed using a standardized, validated CVR quantification pipeline incorporating motion correction, physiological noise regression, and voxelwise modeling of the BOLD signal in response to the vasoactive stimulus.

Control Strategy: Historical Comparison Given the exploratory and interventional nature of this study, a randomized control group is not feasible within this pilot phase. Instead, a historical control cohort will be utilized to contextualize observed changes in BOLD-CVR following lumbar drainage.

The historical cohort includes previously scanned acute ischemic stroke patients with HF2 profiles who underwent BOLD-CVR MRI at two time points (typically 3-7 days apart) but without any interventional procedure between scans. These patients were matched for age, vascular risk factors, infarct location, and NIHSS at baseline.

This allows for a comparison of temporal BOLD-CVR changes occurring naturally in similar patients, thereby enabling preliminary inference about the causal effect of CSF drainage on CVR dynamics.

Outcome Measures

Primary Endpoint:

Change in mean hemispheric and/or MCA-territory BOLD-CVR between pre- and post-drainage imaging.

Secondary Endpoints:

Incidence of adverse events related to lumbar drain (e.g., headache, infection, CSF leak).

Change in NIHSS from baseline to discharge.

Change in mRS at 3-month follow-up.

Incidence of recurrent ischemic stroke within 90 days.

Statistical and Analytical Considerations Given the exploratory nature of this pilot study, no formal power calculation has been performed. However, a target sample size of 10-15 interventional cases has been selected based on feasibility and expected enrollment rates.

Statistical approach:

Pre/post comparisons will be performed using paired statistical tests (e.g., Wilcoxon signed-rank or paired t-test depending on normality) to evaluate changes in BOLD-CVR.

The historical cohort (n ≈ 20-30) will serve as a reference distribution. Between-group comparisons will use mixed-effects models or ANCOVA adjusting for baseline CVR and time between scans.

Exploratory ROC and AUC analyses will be conducted to evaluate whether baseline CVR thresholds predict benefit from CSF drainage.

Adverse event rates and tolerability measures will be reported descriptively.

Missing data will be handled using appropriate methods (e.g., multiple imputation or last observation carried forward), depending on extent and distribution.

Technical Considerations BOLD-CVR acquisition will use echo-planar imaging sequences optimized for T2*-sensitivity, with whole-brain coverage and temporal resolution ≤2s.

Stimulus control will be ensured via synchronized end-tidal gas monitoring or standardized breath-hold timing via visual cueing.

Data analysis will include use of validated toolboxes (e.g., FSL, AFNI, or custom MATLAB pipelines), including individual voxel z-scoring and spatial normalization to MNI space.

Quality control metrics (e.g., framewise displacement, temporal signal-to-noise ratio) will be logged to assess scan integrity.

All scans will be independently reviewed by a neuroradiologist and a neuroimaging researcher.

Data Handling and Ethics All study data will be pseudonymized and stored on secure hospital servers with limited access. BOLD-CVR imaging data, drain parameters, clinical metrics, and safety events will be recorded in a pre-defined electronic case report form (eCRF). Monitoring will be performed according to ICH-GCP principles. This study has been submitted for ethical approval to the responsible Cantonal Ethics Committee (KEK) and notified to Swissmedic as a Category B interventional clinical trial.

Informed consent will be obtained prior to inclusion. For patients lacking decision-making capacity, legal proxy consent will be used, followed by re-consent as soon as feasible. Participation can be withdrawn at any time, and imaging or data will be excluded upon request.

Anticipated Impact This study provides a first step toward evaluating an innovative, low-risk intervention in a high-risk stroke population for whom current treatments are insufficient. If successful, lumbar drainage could become a temporary, targeted approach to improve cerebral perfusion and reduce recurrence risk in patients with exhausted autoregulatory capacity.

The study is expected to yield mechanistic insights and generate effect size estimates to inform a future randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients > 18 years old
* Acute ischemic stroke related to a new uni- or bilateral occlusion of the ICA, MCA (M1- and or M2 segment) or both
* Persisting vascular pathology after the initial treatment.
* Hemodynamic impairment on the BOLD-CVR done within 48 hours after stroke onset.
* Capable of providing informed consent as documented by signature, or if unable, the next of kin (legally authorized representative) must be available for medical decision-making.

Exclusion Criteria:

* Inclusion in any other running scientific study
* Contraindications for MRI, including but not limited to:

  o Pacemakers, metallic implants/prostheses, metallic tattoo dyes.
* Severe glaucoma.
* Unwillingness or inability to perform breathing maneuvers required for BOLD-CVR assessment.
* Major cardiopulmonary diseases, including:

  * Severe uncontrolled asthma bronchiale.
  * Severe chronic obstructive pulmonary disease (COPD, GOLD Stage >2).
  * Diffuse interstitial lung disease.
  * Recent myocardial infarction (acute/subacute).
  * Severe heart failure (NYHA class >2).
* Symptomatic increased intracranial pressure (ICP) or related conditions:

  * Absent/compressed basal cisterns.
  * Compression or displacement of the fourth ventricle.
  * Cerebellar tonsillar herniation (>5mm below the foramen magnum) on initial CT/MRI or on MRI at Day 1.
* Obstructive hydrocephalus, including:

  * Aqueductal stenosis.
  * Enlarged lateral and third ventricles with a normal fourth ventricle.
* Presence of intracranial hemorrhage class >1 (per Heidelberg classification).
* Unilateral or bilateral subdural hematomas.
* Malignant infarction syndrome (supratentorial or infratentorial).
* Decreased level of consciousness at enrollment, not due to aphasia
* New-onset seizures after stroke onset.
* Extensive lumbar surgery history.
* Local or systemic infection:
* Infection at the lumbar drain insertion site.
* Systemic infection at the time of enrollment.
* Severe coagulopathy, including:

  * Moderate/severe thrombocytopenia (<100,000 platelets/µL).
  * Hemophilia or other coagulation disorders.
  * Use of anticoagulants (except for platelet aggregation inhibitors) that cannot be stopped.
  * Within 24 hours after intravenous thrombolysis
* Structural spinal abnormalities, including:

  * Spina bifida.
  * Scoliosis affecting lumbar puncture feasibility.
* Pregnant (confirmed or verbally suspected) or lactating women.
* Inability to follow the procedures of the study, including but not limited to:

  * Severe cognitive impairment (e.g., dementia).
  * Psychiatric disorders affecting cooperation.
  * Severe language barriers preventing study compliance.
* Failure to insert the lumbar drain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in BOLD-CVR Between Pre- and Post-CSF Drainage | From baseline MRI (prior to CSF drainage) to follow-up MRI within 24 hours after completion of drainage (total approx. 2-3days post-enrollment)
  This outcome measures the change in cerebrovascular reactivity (CVR) based on BOLD-MRI performed before and after continuous cerebrospinal fluid (CSF) drainage via lumbar drain. CVR will be quantified as the mean signal response in both the affected hemisphere and the MCA territory during a standardized hypercapnic stimulus (e.g., breath-hold or controlled CO₂). Change will be assessed using validated voxelwise analysis pipelines to determine whether CSF drainage improves impaired vascular reserve in patients with hemodynamic failure. Each patient serves as their own control for evaluating the physiological impact of the intervention.
Change in BOLD-CVR Between Pre- and Post-CSF Drainage | From baseline MRI (prior to CSF drainage) to follow-up MRI within 24 hours after completion of drainage (total approx. 2-3 days post-enrollment)
  This outcome measures the change in cerebrovascular reactivity (CVR) based on BOLD-MRI performed before and after continuous cerebrospinal fluid (CSF) drainage via lumbar drain. CVR will be quantified as the mean signal response in both the affected hemisphere and the MCA territory during a standardized hypercapnic stimulus (e.g., breath-hold or controlled CO₂). Change will be assessed using validated voxelwise analysis pipelines to determine whether CSF drainage improves impaired vascular reserve in patients with hemodynamic failure. Each patient serves as their own control for evaluating the physiological impact of the intervention.

SECONDARY OUTCOMES:
Comparison of BOLD-CVR Change Between Intervention Group and Historical Control Cohort | From baseline MRI (day 0) to follow-up MRI (day 2-3) in both intervention and historical control cohorts
  This outcome evaluates whether the longitudinal change in cerebrovascular reactivity (CVR), as measured by serial BOLD-CVR MRI, differs between patients with acute stroke undergoing lumbar CSF drainage and a matched historical cohort that did not receive the intervention. Patients will be matched based on age, infarct location, and initial hemodynamic status. This comparison will help determine whether observed improvements in CVR exceed natural variability.
Immediate Hemodynamic Impact of Acute CSF Withdrawal on BOLD-CVR | Second BOLD-CVR performed within 30 minutes after post-drainage MRI (typically day 2)
  To assess whether an acute 20 mL CSF removal leads to measurable changes in CVR, BOLD-CVR will be performed twice in rapid succession: once after the standard post-drainage scan and again immediately after CSF extraction. This sequential imaging captures dynamic cerebrovascular reactivity in response to sudden reduction in intracranial pressure.
Incidence of Recurrent Ischemic Stroke | From study enrollment to 90 days post-stroke
  To assess the rate of recurrent ischemic stroke within the study population during the first 90 days following the initial event. An event rate of approximately 40% is expected if the null hypothesis holds. Diagnosis will be confirmed by clinical assessment and imaging (CT or MRI).
Incidence of Lumbar Drain-Related Complications | From drain placement to 7 days post-removal or hospital discharge, whichever occurs later
  To evaluate the safety of lumbar drain placement by assessing procedure-related complications including headache, infection, CSF leakage, hemorrhage, or neurological deterioration. Adverse events will be recorded and categorized by severity and relatedness to the intervention.
Hemodynamic Parameters Associated With Lumbar Drainage | From baseline (pre-drainage) to 48 hours post-drainage completion
  To assess changes in physiological variables before and after lumbar drainage, including mean arterial pressure (MAP), intracranial pressure (ICP), and estimated cerebral perfusion pressure (CPP). These will be measured using non-invasive and/or invasive monitoring techniques.
Neurological and Functional Outcomes at 3 Months as measured using the To evaluate clinical recovery after intervention using the National Institutes of Health Stroke Scale. | From admission to 3-month outpatient follow-up
  To evaluate clinical recovery after intervention using the National Institutes of Health Stroke Scale (NIHSS; score range: 0 to 42, where lower scores indicate less severe neurological impairment), compared to NIHSS scores obtained at admission and early post-drainage time points.
  The NIHSS is composed of 15 items evaluating specific neurological domains-including level of consciousness, gaze, visual fields, motor function (arms and legs), limb ataxia, sensory function, language, speech, and neglect. Each item is scored individually and then summed to produce the total NIHSS score, which reflects the overall severity of the stroke-related neurological deficit.
Functional Outcome in Patients with Acute Ischemic Stroke After the Intervention, as Measured by the Modified Rankin Scale | From admission to 3-month outpatient follow-up
  To assess functional outcome at 3 months post-stroke using the modified Rankin Scale (mRS; score range: 0 to 6, where lower scores indicate less disability and greater independence), compared to baseline and early post-drainage functional status.
  The mRS is a clinician-reported global functional scale that rates the degree of disability or dependence in daily activities. The score is based on a structured clinical assessment or interview, often supplemented by collateral history from caregivers. It reflects the patient's overall level of functioning, with 0 representing no symptoms and 6 representing death.

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan HB van Niftrik, MD PhD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date: Approximately 6 months after publication of the primary results End Date: Up to 5 years after publication, or as long as the data remains scientifically relevant and ethically shareable under applicable regulations
Access Criteria: Qualified researchers affiliated with academic, non-profit, or governmental institutions may request access to de-identified individual participant data (IPD) and supporting documents (study protocol, SAP, ICF, CSR, and analytic code) for secondary analyses that are methodologically sound and ethically approved. Requests must include a detailed research proposal, data use agreement, and evidence of appropriate institutional review. Data will be shared via secure transfer platforms following approval by the study sponsor and/or principal investigator. Commercial entities may be considered on a case-by-case basis if the proposed use aligns with the scientific and ethical goals of the original study.